CLINICAL TRIAL: NCT00924339
Title: The Soy Food Intervention Trial (SOY FIT) for the Treatment of Children and Adolescents With Familial Hypercholesterolaemia - Beneficial Effect of a Soy-Substituted Diet Confirmed by Assessment of Urinary Isoflavone Excretion as Compliance Markers
Brief Title: Soy Food Intervention Trial
Acronym: SOYFIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Kurt Widhalm, Division Nutrition and Metabolism, Department of Pediatrics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOYFIT
Record Dates: First submitted 2009-05-28; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Familial Hypercholesterolemia
Keywords: soy protein; familial hypercholesterolaemia; children and adolescents; isoflavones; FH
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Rapeseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapeseed oil (Placebo Comparator): Control-Group (n = 15) : Diet reduced in SFA, modified in fatty acid pattern. Only rapeseed oil should to be used for preparation of the meals (baking, frying, in salad, and as spread.
  Interventions: Dietary Supplement: rapeseed oil
- Soy protein diet (Experimental): Intervention-Group (n = 15): Fat- modified dietary regime and a minimum amount of soy protein: 0,25 g/ kg BW/d
  Interventions: Dietary Supplement: soy protein diet

INTERVENTIONS:
Dietary Supplement: soy protein diet — Intervention-Group (n = 15): Fat- modified dietary regime and a minimum amount of soy protein: 0,25 g/ kg BW/d
  Arms: Soy protein diet
Dietary Supplement: rapeseed oil — Control-Group (n = 15): Diet reduced in SFA, modified in fatty acid pattern. Only rapeseed oil should to be used for preparation of the meals (baking, frying, in salad, and as spread.
  Arms: Rapeseed oil

SUMMARY:
Familial hypercholesterolemia (FH MIM#143890), an inherited disorder of lipoprotein metabolism, is a risk for early cardiovascular disease (CVD). This autosomal dominant disease is characterized by markedly elevated plasma concentrations of low density lipoprotein (LDL) and total cholesterol (TC), typically well above the 95th percentile for age and sex (1). A defective gene for the LDL-receptor is inherited from one parent (2). The disorder was first noted by Müller in 1939, including familial clustering of tendon xanthomas, high serum cholesterol and early MIs (3).

The present study aims: a) to strengthen the evidence for the hypocholesterolaemic effect of soy protein in children and adolescents affected with FH b) to monitor the compliance of soy consumption as a possible causal factor linked to the variable lipaemic response observed in the previous study c) to assess certain safety markers of soy food consumption (hormone status, thyroid function, bone metabolism) 4) to monitor the adherence to the soy intervention additionally comprise collections of blood and urine samples.

Hypothesis 1: Soya protein-substituted diets change total and LDL-cholesterol, Apolipoprotein B and uric acid serum concentrations.

Primary parameters: Blood analysis

Hypothesis 2: Children and adolescents with FH, in which the cholesterol, LDL-lipoprotein and Apolipoprotein B concentration is not influenced by means of soy protein substituted diet - is it because of a) the effect of non-responder? or b) subjects, who have no regularly dietary soya intake.

Secondary parameters: isoflavones daidzein, glycetein, genistein and equol in the urine samples

DETAILED DESCRIPTION:
The pilot study will include 30 children and adolescents with heterozygous Familial Hypercholesterolemia. All children and adolescents will be recruited from the Paediatrics Outpatient Department of the Division of Clinical Nutrition and Metabolism at the Vienna University Hospital. Furthermore, children of patients with heart stroke, patients from other paediatrics and patients from other children hospitals will be recruited. Inclusion criteria: To be eligible the study participants will have to be aged between 4 and 18 years, do not regularly eat soy food and do not have a protein allergy. The participants are recruited by their familial history and/or their cholesterol levels (elevated over 130 mg/dl and total cholesterol elevated over 200 mg/dl) according to American Academy of Paediatrics criteria. Furthermore they should keep a 7-day nutrition record at the beginning of study. Exclusion criteria: Patients younger than 4 years and older than 18 years, children who are extremely underweight according to Kromeyer Hausschild´s criteria. Children and adolescents with mental disability and with simultaneous medication and protein allergy. Complete physical information will be done and a thorough medical history will be taken in all participants. Physical examination and blood sampling will be performed in the outpatient clinic setting as done routinely.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible the study participants will have to be aged between 4 and 18 years,
* do not regularly eat soy food and do not have a protein allergy.
* the participants are recruited by their familial history and/or their cholesterol levels (elevated over 130 mg/dl and total cholesterol elevated over 200 mg/dl) according to American Academy of Paediatrics criteria

Exclusion Criteria:

* Patients younger than 4 years and older than 18 years,
* children who are extremely underweight according to Kromeyer Hausschild´s criteria.
* Children and adolescents with mental disability and with simultaneous medication and protein allergy.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Blood analysis include: TC, LDLc, HDLc, TG, Lp(a), ApoA1, Apo B, Electrolytes, Albumin, Creatinin and CRP | done in Phase 1: 1st week, Phase 2: 7th week, Phase 3: 13th week

SECONDARY OUTCOMES:
uric acid and the isoflavones: daidzein, glycetein, genistein and equol | done in Phase 1: 1st week, Phase 2: 3rd, 5th, 7th, 9th, 11th week, Phase 3: 13th week

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Nutrition and Metabolism, Department of Pediatrics, Medical University of Vienna, Vienna, Vienna, Austria